CLINICAL TRIAL: NCT05624528
Title: A Double-Blind, Randomized, Placebo-Controlled Study of Tolcapone for OCD
Brief Title: A Clinical Trial of Tolcapone in Obsessive Compulsive Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB22-1729
Record Dates: First submitted 2022-11-14; First posted 2022-11-22 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-06

CONDITIONS: Obsessive-Compulsive Disorder; OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Tolcapone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tolcapone (Experimental): 100mg of tolcapone twice daily for two weeks, then 200mg tolcapone twice daily for the remaining six weeks.
  Interventions: Drug: Tolcapone
- Placebo (Placebo Comparator): 100mg of placebo twice daily for two weeks, then 200mg of placebo twice daily for the remaining six weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tolcapone — catechol-O-methyl transferase inhibitor
  Other Names: Tasmar
  Arms: Tolcapone
Drug: Placebo — Pill that contains no medicine
  Arms: Placebo

SUMMARY:
The primary aim of the present study is to examine the efficacy and safety of tolcapone in adults with moderate to severe OCD.

DETAILED DESCRIPTION:
Based on the mechanism of action and our previous pilot data, the primary aim of the present study is to examine the efficacy and safety of 8-week treatment with tolcapone vs. placebo in adults with moderate to severe OCD, as indicated by a score of at least 21 on the Yale Brown Obsessive Compulsive Scale (YBOCS), a scale of illness severity, at the baseline visit. We hypothesize that tolcapone will significantly improve symptoms of OCD compared to placebo.

A secondary aim of the proposed study is to examine the cognitive effects of tolcapone in OCD, by conducting objective neuropsychological tasks pre- and post-pharmacological trial. The rationale for this approach is that: dopamine plays a key role in cognition; cognitive effects of tolcapone are likely to be relevant in explaining symptomatic effects; and cognitive dysfunction constitutes an important treatment target in OCD that is not generally ameliorated by current first-line interventions. We hypothesize that any symptomatic benefit with tolcapone would also be associated with improvement in executive functions including cognitive flexibility.

Another secondary aim of the proposed study is to evaluate whether the single nucleotide polymorphism (SNP) Val-158-Met polymorphism significantly relates to changes in symptoms and cognition observed with tolcapone. Prior data indicate cognitive effects of tolcapone are affected by this SNP. We hypothesize that the val/val COMT variant will be associated with significantly higher tolcapone-related improvements in cognition and symptoms, since this is linked to lower cortical dopamine function.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 18-65 years
2. Primary diagnosis of OCD
3. YBOCS score of at least 21 at baseline (moderate or higher severity)
4. Ability to understand and sign the consent form

Exclusion Criteria:

1. Unstable medical illness based on history or clinically significant abnormalities on baseline physical examination
2. Current pregnancy or lactation, or inadequate contraception in women of childbearing potential
3. Subjects considered an immediate suicide risk based on the Columbia Suicide Severity rating Scale (C-SSRS) (www.cssrs.columbia.edu/docs)
4. History of psychosis or bipolar disorder based on DSM-5 criteria
5. Alcohol/substance use disorder and/or illegal substance use based on urine toxicology
6. Initiation of psychological interventions within 3 months of screening (those who are continuing with CBT will be included)
7. Use of any new psychotropic medication within 3 months of study entry (stable doses of psychotropics will be allowed)
8. Major cognitive impairment that interferes with the capacity to understand and self-administer medication or provide written informed consent
9. Abnormal liver function tests at baseline
10. MADRS >30 at baseline

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Yale Brown Obsessive Compulsive Scale (YBOCS) | Baseline to Week 8
  A measure of OCD illness severity

SECONDARY OUTCOMES:
CANTAB Cognitive Testing | Baseline to Week 8
  Neuropsychological tasks that measure cognition
Val-158-Met polymorphism | Baseline to Week 8
  Evaluating whether the single nucleotide polymorphism (SNP) Val-158-Met polymorphism significantly relates to changes in symptoms and cognition observed with tolcapone.
Quality of Life Inventory | Baseline to Week 8
  A self-report measure assessing perceived quality of life.
Montgomery-Asberg Depression Rating Scale | Baseline to Week 8
  A 10-item clinical rated scale measuring depression severity.

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Grant, MD, JD, MPH, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No